CLINICAL TRIAL: NCT03887533
Title: Combined Intrathecal and Intravenous VTS-270 Therapy for Liver and Neurological Disease Associated With Niemann-Pick Disease, Type C1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment was poor due to COVID-19 pandemic
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190028; 19-CH-0028
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-10

CONDITIONS: Niemann-Pick Disease, Type C1
Keywords: 2-Hydroxypropyl-B-Cyclodextrin
MeSH Terms: conditions — Niemann-Pick Disease, Type C

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VTS-270 at 500 mg/kg (Experimental): Participant received dose of 500 mg/kg of intravenous VTS-270 administered over 2 hours monthly for 12 months. Participant also received 900 mg intrathecal VTS-270 therapy monthly for 18 months.
  Interventions: Drug: VTS-270
- VTS-270 at 1000 mg/kg (Experimental): Participant received 1000 mg/kg of intravenous VTS-270 over 4 hours monthly for 12 months. Participant also received 900 mg intrathecal VTS-270 therapy monthly for 18 months.
  Interventions: Drug: VTS-270

INTERVENTIONS:
Drug: VTS-270 — Intravenous VTS-270 was administered on a monthly dosing schedule for 12 months. Each participant received one of two doses (500 or 1000mg/kg). Participants also received monthly 900 mg intrathecal VTS-270 therapy.

SUMMARY:
Background:

For people who have Niemann-Pick disease, type C1 (NPC1), cholesterol and other fats have trouble moving out of liver and other tissue cells. This makes the cells sick. Researchers want to find out if a drug called VTS-270 can help.

Objective:

To test if VTS-270 is safe and effective in treating chronic liver disease associated with NPC1.

Eligibility:

People ages 3-60 with NPC1

Design:

Participants may be screened by phone or under another protocol.

Participants will have visits once a month for 12 months. If they have intrathecal injections, the study may last 15 months or more. The first visit will last about 5 days. Others will last 2-3 days.

Participants will get VTS-270 injected into a vein at each visit. They can also choose to have intrathecal injections. These are like spinal taps.

Some visits will also include:

Physical exam

Urine tests

Blood tests. A small tube or needle will be inserted into the participants vein to collect blood. The small tube will also be used to give the VTS-270.

Hearing tests: For one test, participants will have electrodes taped to their head. These will record brain waves.

Breathing tests

Ultrasound of abdomen: Sounds waves will take pictures of the participant s body.

Chest x-ray: This is a picture of the lungs.

DETAILED DESCRIPTION:
Niemann-Pick disease type C (NPC) is a lethal, autosomal recessive, lysosomal storage disorder characterized by neurodegeneration in early childhood and death in adolescence. NPC results from mutation of either the NPC1 (approximately 95% of cases) or NPC2 genes. Biochemically, NPC is characterized by the endolysosomal storage of unesterified cholesterol and lipids in both the central nervous system and peripheral tissues such as the liver. Individuals with NPC demonstrate progressive cerebellar ataxia and dementia. Acute cholestatic liver disease is frequently observed in the neonatal/infantile period but subsequently resolves. However, chronic, sub-clinical liver disease persists. Intrathecal 2-hydroxypropyl-beta-cyclodextrin (HPbetaCD, VTS-270) has proven effective in reducing signs and prolonging life in NPC1 animal models, and Phase 1/2a data support efficacy in NPC1 patients. Parenteral administration of VTS-270 has also been shown to be effective in treating liver disease in the NPC1 cat.

In this Phase 1/2a, open-label, randomized, parallel dose, single-center study, we will examine whether VTS-270 can be used to treat chronic subacute liver disease in NPC1 patients. Our primary objective is to determine the safety and tolerability of intravenous VTS-270 in NPC1 disease. Secondary objectives will be to evaluate the efficacy of VTS-270 to reduce plasma cholestane-3beta,5alpha,6beta-triol, an NPC1-specific pharmacodynamic biomarker, and to normalize the degree of liver injury. Exploratory testing will include lipid and protein biomarkers. This study will evaluate three dose levels (500, 1000 and 1500 mg/kg) administered monthly for twelve months. Safety will be assessed by adverse event recording, clinical laboratory testing and physical examination. Clinical efficacy will be evaluated by assessment of liver chemistries, determination of liver size; and liver STIFFNESS. Biochemical efficacy will be assessed by measurement of plasma cholestane-3beta,5alpha,6beta-triol and other biomarkers.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age greater than or equal to 3 and less than or equal to 60 years old at time of enrollment
2. Diagnosis of NPC1 based upon one of the following:

   A. Two NPC1 mutations

   B. Biochemical Positive for NPC (oxysterol/bile acid and sphingomyelinase levels consistent with a diagnosis of NPC) and one NPC1 mutation
   * NPC1 mutations will be interpreted using standards established for the interpretation of sequence variants [33].
   * Oxysterol/Bile Acid testing refers to cholestane-3beta,5 ,6beta-triol [7, 8] or 3beta,5alpha,6beta-trihydroxycholanic acid and its glycine conjugate [34].
3. Evidence of NPC1-related liver disease as defined by one of the following:

A. Abnormal liver chemistries as defined by one of the following:

i. Plasma aspartate aminotransferase (AST) greater than or equal to 1.5-times age-appropriate upper limit of normal

ii. Plasma aspartate aminotransferase (AST) greater than or equal to 1.25-times age-appropriate upper limit of normal and plasma alanine aminotransferase (ALT) > 1.25-times age-appropriate upper limit of normal

iii. Plasma aspartate aminotransferase (AST) greater than or equal to 1.25-times age-appropriate upper limit of normal and AST/ALT ratio greater than or equal to 2.0 AND Abnormal liver chemistries as defined above at least 8 weeks apart.

B. Abnormal Liver Ultrasound* defined as one of the following:

1. Intraparenchymal echogenic bands consistent with fibrosis
2. Abnormal liver echogenicity with AST or ALT above the upper limit of normal.
3. Hepatomegaly with AST or ALT above the upper limit of normal.

   To define hepatomegaly, we will use the suggested limit of normal of the longitudinal dimension of the right lobe of the liver. These values are approximately 2 standard deviations above the mean.

   C. Abnormal liver stiffness (FibroScan**) for age.

   To define Liver Stiffness Measurement we will use the normal age dependent ranges. Values above the 95th centile will be considered abnormal.
4. Ability to travel to the NIH Clinical Center repeatedly for evaluation and follow-up.
5. Willingness to discontinue all non-prescription supplements, except for an age-appropriate multivitamin/mineral supplement.
6. Stable miglustat dose for 3 months prior to entry into the IV portion of the trial.
7. Women of reproductive age must be willing to use an effective method of contraception for the duration of the trial if sexually active.
8. Willingness to participate in all aspects of the IV trial

EXCLUSION CRITERIA:

* Age <3 or > 60 years of age at time of enrollment in the trial.
* Subjects who have received any form of parenteral cyclodextrin, an HDAC inhibitor, or an experimental therapy for NPC in the prior six months. Prior Intrathecal VTS-270 treatment is allowed.
* History of hypersensitivity reactions to cyclodextrin or components of the formulation.
* Pregnancy or breastfeeding. Females of childbearing potential unwilling to utilize a highly effective form of contraception (i.e., barrier method with spermicide, intrauterine device, steroidal contraceptive in conjunction with a barrier method, or abstinence if it is the patient s baseline preference) for the duration of the study and for 30 days after participation.
* Any systemic infection at the time of enrollment.
* Neutropenia, defined as an absolute neutrophil count (ANC) of less than 1,500 per microliter. Subjects with benign cyclic/ethnic neutropenia may be enrolled if not clinically symptomatic.
* Thrombocytopenia defined as a platelet count less than 75,000 per microliter.
* Established history of a chronic clotting or bleeding disorder.
* Use of anticoagulants within 3 months of enrollment
* Severe or acute liver disease as defined by one of the following:

A. AST or ALT greater than 10-times age-appropriate upper limit of normal

B. Jaundice or right upper quadrant pain

C. International Normalized Ratio (INR) >1.8

* Individuals with AST and ALT greater than 4-times the age-appropriate upper limit of normal will be excluded if they have a positive NIH Clinical Center Viral Markers Hepatitis Screen (HBsAG, anti-HCV and Anti-HAV IgM). This screening test will not be obtained unless AST and ALT are elevated. An equivalent panel from another laboratory may be used if this elevation is noted on screening. Individuals excluded under this criterion may be rescreened after the acute pathology resolves (e.g. Hepatitis A infection).
* Presence of anemia defined as two standard deviations below normal for age and gender.
* Serum creatinine level greater than 1.5 times the age-appropriate upper limit of normal OR FOR INDIVIDUALS >= 6 years of age an eGRF < 60 mL/min 1.73 m squared
* Hematuria on a single urinalysis, as defined by the American Urological Association (AUA) as five or more red blood cells per high-power field on microscopic evaluation of urinary sediment from a properly collected urinalysis specimen. The patient will not be excluded if two subsequent urine specimens are negative for hematuria as defined by the AUA.
* Proteinuria (1+ protein on repeat urinalysis) unless evaluated and classified as benign.
* Active pulmonary disease, oxygen requirement or clinically significant history of decreased blood oxygen saturation (SaO2 <95% on room air), pulmonary therapy, daily use of a cough assist device or pulmonary vest, requiring active suction, or with a tracheostomy.
* Patients with uncontrolled seizures per either of the criteria below.

  1. Unstable frequency, type or duration of seizures. Quantified by a seizure log over one month prior to enrollment.
  2. Subject requiring antiepileptic medication changes (other than dose adjustments for weight) in the month prior to enrollment.
* Individuals receiving parenteral nutrition will be excluded.
* Patients, who in the opinion of the investigators, are unable to comply with the protocol or have specific health concerns that would potentially increase the risk of participation.

Additional exclusion criteria for intrathecal VTS-270

1. Neurologically asymptomatic. Determination made by the investigators based on history, neurological exam and consultant input.
2. Suspected infection of the central nervous system
3. Spinal deformity that would impact the ability to perform a lumbar puncture
4. Skin infection in the lumbar region
5. Prior use of anticoagulants or a bleeding disorder with increased risk of clinical bleeding.
6. Patients unable to complete a behavioral audiological evaluation including pure-tone threshold assessment (500 Hz to 8000 Hz). In consultation with the medical monitor and audiologists, a sedated ABR may be utilized to monitor ototoxicity if the participant is being sedated to receive IT VTS-270.
7. Patients, who in the opinion of the investigators, are unable to comply with the protocol or have specific health concerns that would potentially increase the risk of participation.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Vanier MT. Niemann-Pick disease type C. Orphanet J Rare Dis. 2010 Jun 3;5:16. doi: 10.1186/1750-1172-5-16. PMID 20525256
- [Background] Porter FD, Scherrer DE, Lanier MH, Langmade SJ, Molugu V, Gale SE, Olzeski D, Sidhu R, Dietzen DJ, Fu R, Wassif CA, Yanjanin NM, Marso SP, House J, Vite C, Schaffer JE, Ory DS. Cholesterol oxidation products are sensitive and specific blood-based biomarkers for Niemann-Pick C1 disease. Sci Transl Med. 2010 Nov 3;2(56):56ra81. doi: 10.1126/scitranslmed.3001417. PMID 21048217
- [Background] Ory DS, Ottinger EA, Farhat NY, King KA, Jiang X, Weissfeld L, Berry-Kravis E, Davidson CD, Bianconi S, Keener LA, Rao R, Soldatos A, Sidhu R, Walters KA, Xu X, Thurm A, Solomon B, Pavan WJ, Machielse BN, Kao M, Silber SA, McKew JC, Brewer CC, Vite CH, Walkley SU, Austin CP, Porter FD. Intrathecal 2-hydroxypropyl-beta-cyclodextrin decreases neurological disease progression in Niemann-Pick disease, type C1: a non-randomised, open-label, phase 1-2 trial. Lancet. 2017 Oct 14;390(10104):1758-1768. doi: 10.1016/S0140-6736(17)31465-4. Epub 2017 Aug 10. PMID 28803710
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CH-0028.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events by Grade
Description: Adverse events (AEs) were used to determine safety and assess safety of intravenous VTS-270 in subjects with Niemann-Pick Disease, type C1. Assessment of safety was made by evaluation of summary statistics of adverse events and unanticipated problems. AEs were assessed using CTCAE version 5.0 grades 1-5.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL*.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL**.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to AE
Time Frame: 18 months
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants
  Grade 1 | 1 | 1
  Grade 2 | 1 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

2. Primary Outcome: Participants With Reduction in Plasma Cholestane-3β
Description: Efficacy of IV VTS-270 in treating chronic liver disease associated with Niemann-Pick Disease, type C1 as measured by reduction in plasma cholestane-3β, an NPC1-specific pharmacodynamic biomarker
Time Frame: Assessed at baseline and at 52 weeks
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

3. Primary Outcome: Participants With Reduction in Plasma Bile Acid B (5α)
Description: Efficacy of IV VTS-270 in treating chronic liver disease associated with Niemann-Pick Disease, type C1 as measured by reduction in bile acid B (5α), an NPC1-specific pharmacodynamic biomarker
Time Frame: Assessed at baseline and at 52 weeks
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

4. Primary Outcome: Participants With Reduction in C-Triol (6β-triol)
Description: Efficacy of IV VTS-270 in treating chronic liver disease associated with Niemann-Pick Disease, type C1 as measured by reduction in C-Triol (6β-triol), an NPC1-specific pharmacodynamic biomarker
Time Frame: Assessed at baseline and at 52 weeks
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

5. Secondary Outcome: Participants With Reduction in Liver Stiffness (kPa)
Description: Efficacy of IV VTS-270 in treating chronic liver disease associated with Niemann-Pick Disease, type C1 as measured by reduction in liver stiffness (kPa)
Time Frame: Assessed at baseline and at 52 weeks
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

6. Secondary Outcome: Participants With Reduction in Alanine Aminotransferase Level
Description: Efficacy of IV VTS-270 in treating chronic liver disease associated with Niemann-Pick Disease, type C1 as measured by reduction of serum alanine aminotransferase level (ALT)
Time Frame: Assessed at baseline and at 52 weeks
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

7. Secondary Outcome: Participants With Reduction in Aspartate Aminotransferase
Description: Efficacy of IV VTS-270 in treating chronic liver disease associated with Niemann-Pick Disease, type C1 as measured by reduction of serum aspartate aminotransferase (AST) level
Time Frame: Assessed at baseline and at 52 weeks
Population: All participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | VTS-270 at 500 mg/kg | VTS-270 at 1000 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTS-270 at 500 mg/kg (N=1) | VTS-270 at 1000 mg/kg (N=1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTS-270 at 500 mg/kg (N=1) | VTS-270 at 1000 mg/kg (N=1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Cardiac disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Activated partial thromboplastin time (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Haematuria (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was poor due to COVID-19 pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03887533/Prot_SAP_000.pdf